CLINICAL TRIAL: NCT04558281
Title: Continuous Erector Spinae Plane Blocks for Analgesia and Improving Incentive Spirometry Following Traumatic Rib Fractures
Brief Title: Continuous Erector Spinae Plane Blocks for Rib Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Could only enroll 4 subjects in nearly 2 years
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor in Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cESPB for Rib Fractures
Record Dates: First submitted 2020-09-13; First posted 2020-09-22 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Rib Fractures; Trauma; Anesthesia; Anesthesia, Local
MeSH Terms: conditions — Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, placebo-controlled, parallel group clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study solution containing either local anesthetic (ropivacaine) or saline will be prepared by the UCSD Investigational Drug Study Service. Both ropivacaine and normal saline are clear and indistinguishable visually.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): This group will receive a single injection nerve block of ropivacaine 0.5% (20 mL) followed by an infusion/boluses of ropivacaine 0.3% (continuous block)
  Interventions: Drug: Active ropivacaine 0.3% erector spinae plane perineural administration
- Placebo (Placebo Comparator): This group will receive a single injection nerve block of ropivacaine 0.5% (20 mL) followed by an infusion/boluses of normal saline
  Interventions: Drug: Placebo erector spinae plane perineural administration

INTERVENTIONS:
Drug: Active ropivacaine 0.3% erector spinae plane perineural administration — Ropivacaine 0.3% administration via an erector spinae plane perineural catheter
  Arms: Active Treatment
Drug: Placebo erector spinae plane perineural administration — Normal saline administration via an erector spinae plane perineural catheter
  Arms: Placebo

SUMMARY:
Rib fractures are one of the most common injuries in trauma patients. These fractures are associated with significant pain as well as decreased ability to inspire deeply or cough to clear secretions, which together lead to complications of the lungs and breathing which leads to risks of further injury and even death.

One recent study found that the ability to move air into and out of the lungs practically doubled with the administration of a single-injection Erector Spainae Plane Block (ESPB) while pain levels nearly halved. However, a single-injection nerve block lasts less than 24 hours while a perineural local anesthetic infusion (also termed a "continuous peripheral nerve block") may be administered for multiple days. This entails inserting a tiny tube through the skin and into the area around the nerves, after which more local anesthetic may be administered prolonging the numbing effects.

The possibility of extending the duration of a ESPB with local anesthetic administration via a perineural catheter has not be investigated. We therefore are conducting a randomized, triple-masked, placebo-controlled, parallel-arm study to investigate the addition of a continuous ESPB to a single-injection ESPB following traumatic rib fractures.

The primary outcome of this study will be the maximum inspired volume measured by incentive spirometry on the afternoon following the nerve block procedure. We hypothesize that the maximum inspired volume will be significantly increased in the afternoon following the procedure with the addition of a continuous ESPB to a single-injection ESPB.

DETAILED DESCRIPTION:
Rib fractures are one of the most common injuries in trauma patients. These fractures are associated with significant pain as well as decreased ability to inspire deeply or cough to clear secretions, which together lead to complications of the lungs and breathing which leads to risks of further injury and even death.

The erector spinae plane block (ESPB) is a nerve block that covers multiple rib fractures with a single injection. This block entails injecting local anesthetic in the back superficial to the vertebral bodies. One study found that the ability to move air into and out of the lungs practically doubled with the administration of a single-injection ESPB while pain levels nearly halved.

A single-injection nerve block lasts less than 24 hours while a perineural local anesthetic infusion (also termed a "continuous peripheral nerve block") may be administered for multiple days. This entails inserting a tiny tube through the skin and into the area around the nerves, after which more local anesthetic may be administered prolonging the numbing effects. The possibility of extending the duration of a ESPB with local anesthetic administration via a perineural catheter has not be investigated.

We therefore are conducting a randomized, tripe-masked, placebo-controlled, parallel-arm study to investigate the addition of a continuous ESPB to a single-injection ESPB following traumatic rib fracture. Subjects will be individuals who present with rib fracture(s) and significant pain. Those who consent to participate in this study will have an ESP catheter inserted using ultrasound-guidance on the ipsilateral side at the level of the inferior-most fracture. For bilateral fractures, a second catheter will also be inserted on the remaining side. The single-injection ESPB will be administered to each catheter with 20 mL of ropivacaine 0.5% (with epinephrine).

Subjects with an accurately-inserted catheter based on visualization of local anesthetic spread will be allocated to one of two possible perineural treatments stratified by unilateral vs. bilateral fractures (1:1 ratio in blocks of 2):

1. active (ropivacaine 0.3%)
2. placebo (normal saline)

Computer-generated randomization lists will be created by the UCSD Investigational Drug Service which will keep the randomization lists and not release them to the investigators until the study is completed, at which time they will provide lists of subjects who received "Treatment A" and "Treatment B" so that the statistician can analyze the data. Only after the analysis is complete will "Treatment A" and "Treatment B" be defined for the investigators for manuscript preparation [producing a triple-masked study]. Of note, for bilateral catheters the treatments on both sides will always be identical: each subject will be randomized to a single treatment and not each side of bilateral cases.

Subjects will receive a basal infusion of study fluid (ropivacaine vs. placebo) 1 mL/h to keep the catheter lumen patent as soon as the infusion pump is initiated with a 500 mL reservoir. In addition, intermittent boluses (13 mL programmed automatic bolus every 2 hours) will begin 5 hours after pump initiation. For bilateral catheters, a 6-hour delay for one of the pumps will ensure that the pair of pumps alternate sides for the bolus doses each hour. This protocol will provide nearly 71-72 hours of study fluid administration.

Following local anesthetic reservoir exhaustion, subjects or their caretakers will remove the catheters with instructions provided by phone. This is standard at UC San Diego for all ambulatory continuous peripheral nerve blocks and will not be unique to study participation. The catheter is disposable in the trash and the infusion pump will be returned using a pre-addressed and postage-paid envelope provided to subjects prior to leaving the hospital.

Subjects will be contacted by telephone to collect study data on post procedure days 1, 2, 7, and at months 0.5, 1, 1.5, 2, 3, 6, and 12.

The ultimate objective of the proposed line of research is to determine if the addition of a continuous ESPB to a single-injection ESPB prolongs analgesia following traumatic rib fractures; and, if this analgesic intervention improves pulmonary mechanics measured with incentive spirometry.

Specific Aim 1: To determine if the addition of a continuous ESPB to a single-injection ESPB improves maximum inspiratory volume following traumatic rib fracture(s).

Hypothesis 1a: The maximum inspired volume will be significantly increased in the afternoon following the procedure [primary endpoint] as well as at other time points following the procedure [secondary end points] with the addition of a continuous ESPB to a single-injection ESPB [measured with an incentive spirometer].

Hypothesis 1b: The maximum inspired volume as a percentage of the baseline will be significantly increased in the afternoon following the procedure [secondary endpoint of greatest interest], as well as at other time points following the procedure [secondary end points] with the addition of a continuous ESPB to a single-injection ESPB [measured with an incentive spirometer].

Specific Aim 2: To determine if the addition of a continuous ESPB to a single-injection ESPB decreases the pain associated with rib fracture(s).

Hypothesis 2a: The severity of rib fracture pain at rest will be significantly decreased within the 12 months following the procedure with the addition of a continuous ESPB to a single-injection ESPB [measured using the Numeric Rating Scale for pain].

Hypothesis 2b: The severity of rib fracture pain when using the spirometer or coughing will be significantly decreased within the 12 months following the procedure with the addition of a continuous ESPB to a single-injection ESPB [measured using the Numeric Rating Scale for pain].

Hypothesis 2c: The incidence of chronic rib fracture pain will be significantly decreased 6 and 12 months following a rib fracture with the addition of a continuous ESPB to a single-injection ESPB [measured using the Numeric Rating Scale for pain].

Hypothesis 2d: The severity of chronic rib fracture pain will be significantly decreased 6 and 12 months following a rib fracture with the addition of a continuous ESPB to a single-injection ESPB [measured using the Numeric Rating Scale for pain].

ELIGIBILITY:
Inclusion Criteria:

* having a total of 1-6 rib fractures at least 3 cm distal to the costo-transverse joint (bilateral fractures are acceptable, but the total of the two sides combined must not exceed 6 fractures)
* regional anesthetic requested by the admitting service
* patient accepting of a perineural catheter insertion and subsequent study fluid treatment.

Exclusion Criteria:

* chronic opioid use (daily use within the 2 weeks prior to presentation and duration of use > 4 weeks; of note, any testing for opioid use will not occur as part of the study, but may as standard of care)
* pregnancy
* incarceration
* inability to communicate with the investigators
* weight < 45 kg or morbid obesity (body mass index > 40 kg/m2)
* comorbidity precluding either perineural catheter insertion or subsequent ambulatory perineural local anesthetic administration (e.g., current infection at the catheter insertion site, known hepatic or renal insufficiency, immune-compromised status of any etiology)
* any patient unable to correctly perform incentive spirometry as this is the primary outcome measure
* any patient with any degree of decreased mental capacity as determined by the surgical service
* any reason an investigator believes study participation would not be in the best interest of the potential subject
* flail chest
* chest tube
* fracture of the 1st rib on either side
* any injury other than the rib fracture(s) that potentially effects inspiratory effort or volume (e.g., clavicle fracture)
* inability to contact the investigators during the perineural administration, and vice versa (e.g., lack of telephone access).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Finneran IV, MD, Study Director — University of California, San Diego; Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (3.5) | 40.5 (21.9) | 39.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Height [Mean (Standard Deviation); unit: meters] | 1.8 (0.1) | 1.7 (83.7) | 1.75 (43.2)
Weight [Mean (Standard Deviation); unit: kg] | 83.7 (16.5) | 68.4 (12.1) | 73 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Inspired Volume - Absolute
Description: Measured via a handheld incentive spirometer. The best of three measurements will be recorded as the maximum inspired volume.
Time Frame: Between 1200 and 1700 on the day following the procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
mL | 2500 (707) | 2625 (530)

2. Secondary Outcome: Maximal Inspired Volume - Absolute
Description: as for outcome 1
Time Frame: Afternoons on postoperative days 2 and 7, postoperative months 0.5, 1, 1.5, 2, 3, 6, and 12
Population: At two time points, neither patient in the treatment group could be reached or no longer had the incentive spirometer to produce the measurement.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
mL
  Day 2 | 2375 (1237) | 2500 (707)
  Day 7 | 2750 (707) | 2750 (707)
  Day 14 | 3250 (354) | 3125 (177)
  Month 1 | 3500 (0) | 3250 (0)
  Month 1.5 | 3375 (177) | 3375 (177)
  Month 2 | 3500 (0) | 3625 (177)
  Month 3: number analyzed (Participants) | 0 | 2
  Month 3 |  | 3875 (177)
  Month 6 | 3500 (0) | 4000 (0)
  Month 12: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Maximal Inspired Volume - Percentage Change From Baseline Prior to Intervention
Description: as for outcome 1
Time Frame: Afternoons on postoperative days 1, 2 and 7, postoperative months 0.5, 1, 1.5, 2, 3, 6, and 12
Population: Some patients could not be reached or no longer had their incentive spirometer to measure the outcome
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
percentage change
  Day 1 | 283 (24) | 263 (53)
  Day 2 | 200 (0) | 250 (71)
  Day 7 | 2750 (707) | 2750 (707)
  Day 14 | 375 (35) | 313 (18)
  Month 1 | 3500 (0) | 3250 (0)
  Month 1.5 | 392 (59) | 338 (18)
  Month 2 | 467 (0) | 363 (0)
  Month 3: number analyzed (Participants) | 0 | 2
  Month 3 |  | 388 (18)
  Month 6 | 467 (0) | 400 (0)
  Month 12: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Brief Pain Inventory (Short Form, Interference Subscale)
Description: The Brief Pain Inventory (short form, Interference scale) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning [7 questions related specifically to rib fracture pain and not other injuries]. We calculated the total score of the 7 questions combined. The minimum is zero (no interference, better outcome) and the maximum is 70 (maximum interference, worse outcome).
Time Frame: Months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Month 0.5 | 33 (9.9) | 5 (1.4)
  Month 1 | 2 (2.8) | 1 (1.4)
  Month 1.5 | 8 (11.3) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

5. Secondary Outcome: Rib Fracture Pain When Using an Incentive Spirometer
Description: Pain rated from 0-10 using a Numeric Rating Scale with 0 equivalent to no pain and 10 equivalent to the worst imaginable pain
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Population: Patients could not be reached at all timepoints and therefore data could not be collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | 5.0 (0) | 5 (1.4)
  Day 2 | 6.0 (1.4) | 4.5 (2.1)
  Day 7 | 5 (1.4) | 4 (0)
  Month 0.5 | 3.5 (0.7) | 3 (1.4)
  Month 1 | 0 (0) | 0 (0)
  Month 1.5 | 4 (4.2) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12: number analyzed (Participants) | 1 | 1
  Month 12 | 0 (0) | 0 (0)

6. Secondary Outcome: WORST Rib Fracture Pain in Previous 24 Hours
Description: as for outcome 5
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | 9 (1.4) | 5.8 (2.5)
  Day 2 | 9 (1.4) | 7 (0)
  Day 7 | 7.5 (0.7) | 7 (1.4)
  Month 0.5 | 5 (1.4) | 4 (0)
  Month 1 | 1 (0) | 1 (1.4)
  Month 1.5 | 2 (1.4) | 0.5 (.7)
  Month 2 | 1 (1.4) | 0 (0)
  Month 3 | 1 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

7. Secondary Outcome: AVERAGE Rib Fracture Pain in Previous 24 Hours
Description: as for outcome 5
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | 3.5 (.7) | 4 (2.8)
  Day 2 | 5 (0) | 3.5 (2.1)
  Day 7 | 3 (0) | 4.5 (.7)
  Month 0.5 | 2.5 (.7) | 1.5 (.7)
  Month 1 | 0 (0) | 0.5 (0.7)
  Month 1.5 | .5 (.7) | 0 (0)
  Month 2 | .5 (.7) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

8. Secondary Outcome: LEAST Rib Fracture Pain in Previous 24 Hours
Description: as for outcome 5
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | .5 (.7) | 3 (2.8)
  Day 2 | 1.5 (.7) | 2 (2.8)
  Day 7 | 1 (0) | 3 (1.4)
  Month 0.5 | .5 (.7) | 0 (0)
  Month 1 | 0 (0) | 0 (0)
  Month 1.5 | 0 (0) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

9. Secondary Outcome: CURRENT Rib Fracture Pain in Previous 24 Hours
Description: as for outcome 5
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | 1.5 (21) | 3.5 (3.5)
  Day 2 | 5 (0) | 4 (2.8)
  Day 7 | 3.5 (.7) | 4.5 (.7)
  Month 0.5 | 3.5 (.7) | 1 (0)
  Month 1 | 0 (0) | 0 (0)
  Month 1.5 | 0 (0) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

10. Secondary Outcome: Opioid Consumption
Description: Amount of opioid used in last 24 hours (ultimately measured in morphine equivalents)
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
mg
  Day 1 | 10 (0) | 2.5 (3.5)
  Day 2 | 12.5 (10.6) | 5 (0)
  Day 7 | 10 (7.1) | 2.5 (3.5)
  Month 0.5 | 0 (0) | 0 (0)
  Month 1 | 0 (0) | 0 (0)
  Month 1.5 | 0 (0) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

11. Secondary Outcome: Sleep Disturbances Due to Rib Fracture Pain
Description: Number of awakenings due to rib fracture pain the previous night
Time Frame: Days 1, 2, and 7, and months 0.5, 1, 1.5, 2, 3, 6, 12 following procedure
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 2 | 2
awakenings
  Day 1 | 0.5 (0.7) | 1.0 (1.4)
  Day 2 | 1 (1.4) | 0.5 (0.7)
  Day 7 | .5 (.7) | 1 (0)
  Month 0.5 | 0 (0) | 1. (1.4)
  Month 1 | 0 (0) | 0 (0)
  Month 1.5 | 0 (0) | 0 (0)
  Month 2 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)
  Month 12 | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04558281/Prot_SAP_000.pdf